CLINICAL TRIAL: NCT05147363
Title: Shockwave: Disruption for A Better Fit
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Cardiovascular Institute of the South Clinical Research Corporation (Other)
Collaborators: Shockwave Medical, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: CardiovascularIS
Record Dates: First submitted 2021-10-15; First posted 2021-12-07 (Actual); Last update posted 2021-12-07 (Actual); Status verified 2021-11

CONDITIONS: Peripheral Arterial Disease
MeSH Terms: conditions — Peripheral Arterial Disease

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Shockwave Intravenous lithotripsy with a Supera stent — Pre-dilation with the option of using a 2-3mm balloon to cross a lesion for lithotripsy with the shockwave device followed by placement of supera stent.

SUMMARY:
Recent clinical trial results demonstrate that IVL can increase lumen area by emitting sonic pressure waves, with less inflation pressure as compared to traditional angioplasty balloon dilation and resulting in minimal trauma to the vessel. Therefore, the use of IVL prior to placement of a stent for severely calcified femoral popliteal arteries may be associated with more successful stent implants and better long-term patency, resulting in a decrease in cardiovascular events. The investigator will evaluate the success by defining as lesion stenosis less than 30% and no evidence of Major Adverse Cardiac Event including death or any amputation of the index limb within 30 days of the procedure.

DETAILED DESCRIPTION:
The purpose of this study is to evaluate the immediate and long term effectiveness of using intravenous lithotripsy followed by the placement of a Supera stent for the treatment of calcified femoral popliteal arteries. The use of IVL and Supera stent will be predetermined by the investigator according to inclusion criteria and the need for treatment and stenting combined, will be confirmed through the use of intravascular ultrasound and the investigators judgment for best practice. Following enrollment and index procedure, the subject will be followed prospectively for one year.

ELIGIBILITY:
Inclusion Criteria:

* age ≥ 18 years
* Treatment for de novo, densely calcified femoral popliteal arteries with 70-100% stenosis as measured by IVUS.
* Lesion lengths up to 140 mm.
* Planned follow-up within the health clinic.

Exclusion Criteria:

* Calcified femoral popliteal arteries that show <70% stenosis by angiography.
* Calcified femoral popliteal arteries with 100% stenosis in which the lesion cannot be crossed after pre-dilation with a 2-3mm balloon.
* Unable or unwilling to provide informed consent, including but not limited to cognitive or language barriers (reading or comprehension).
* Thrombophlebitis or deep venous thrombus, within the previous 30 days.
* Evidence of end stage renal disease (ESRD) or stage 5 chronic kidney disease (CKD).
* Currently receiving treatment in an investigational device or drug study or anticipate participating in an investigational device or drug study for the duration of this study.
* Anticipated life expectancy less than 6 months.
* Lack of phone or email for contact.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: 50 consented adults 18 years of age or older, identified to have de novo, severely calcified femoral popliteal arteries requiring revascularization
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2020-12-07 (Actual); Primary Completion 2022-06-07 (Estimated); Study Completion 2022-12-07 (Estimated)

PRIMARY OUTCOMES:
Effectiveness | immediately after the intervention
  determining effectiveness of the procedure will be defined as final residual stenosis of <30% post-stent placement, as measured by IVUS.
Major adverse cardiac events | up to 30 days
  a composite of Major Adverse Cardiac events (MACE) including death and any amputation of the index limb within 30 days. Study success will be defined as those patients who meet both the effectiveness and safety objectives.

SECONDARY OUTCOMES:
increase in minimum lumen area | immediately following intervention
  the change in minimum lumen area following IVL treatment measured in mm2 by intravenous ultrasound
Patency of index vessel | up to 6 months
  primary patency rate of ≥80% measured by extravascular ultrasound
Extended patency of index vessel | 1 year
  long term patency of index vessel of ≥80% measured by extravascular ultrasound
improved ankle-brachial index | 1 year
  an increase in ankle-brachial index measured by the ankle pressure in mmHg divided by the brachial pressure in mmHg

OTHER OUTCOMES:
improved quality of life | 1 year
  relief of symptoms related to intermittent claudication (IC) as reported by the patient during follow up visit

CONTACTS AND LOCATIONS:
Locations (1):
- Cardiovascular Institute of the South, Houma, Louisiana, United States

IPD SHARING:
Plan to Share IPD: No
Individual participant data will be kept within CIS and not shared with anyone outside of the organization